CLINICAL TRIAL: NCT03364491
Title: Tranexamic Acid for the Prevention of Obstetrical Hemorrhage After Cesarean Delivery: A Randomized Controlled Trial
Brief Title: Tranexamic Acid for the Prevention of Obstetrical Hemorrhage After Cesarean
Acronym: TXA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The George Washington University Biostatistics Center (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HD36801-TXA; U10HD036801 (NIH); UG1HD087230 (NIH); UG1HD027869 (NIH); UG1HD040500 (NIH); UG1HD034208 (NIH); UG1HD027915 (NIH); UG1HD040485 (NIH); UG1HD053097 (NIH); UG1HD040544 (NIH); UG1HD040545 (NIH); UG1HD040560 (NIH); UG1HD040512 (NIH); UG1HD087192 (NIH)
Record Dates: First submitted 2017-11-22; First posted 2017-12-06 (Actual); Results first posted 2023-01-19 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Obstetrical Complications; Hemorrhage; Labor and Delivery
Keywords: Tranexamic Acid; Hemorrhage; Cesarean
MeSH Terms: conditions — Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive either TXA (1 gram [10cc] mixed with 40 cc of normal saline) administered intravenously or a placebo control of 50 cc of normal saline administered intravenously
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The patient nor the clinical staff will be aware of the treatment assignment. The TXA or placebo solutions will be prepared by the center research pharmacies.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tranexamic Acid (Experimental): Tranexamic Acid for intravenous administration
  Interventions: Drug: Tranexamic Acid
- Placebo (Placebo Comparator): Normal saline for intravenous administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tranexamic Acid — A single dose of Tranexamic Acid (1 gram) in normal saline for a total of 50cc, administered intravenously immediately following umbilical cord clamping (or as soon as possible afterward)
  Other Names: TXA
  Arms: Tranexamic Acid
Drug: Placebo — 50 cc normal saline administered intravenously immediately following umbilical cord clamping (or as soon as possible afterward)
  Arms: Placebo

SUMMARY:
A randomized placebo-controlled trial of 11,000 women to assess whether tranexamic acid as prophylaxis lowers the risk of postpartum hemorrhage in women undergoing a cesarean delivery.

DETAILED DESCRIPTION:
Obstetrical hemorrhage is a common cause of maternal morbidity and mortality worldwide. The frequency and severity of hemorrhage is significantly higher after cesarean delivery than vaginal delivery. Recent evidence has emerged about the importance of the fibrinolytic pathway in the pathophysiology of hemorrhage in different clinical scenarios including trauma-associated bleeding, cardiovascular surgery, and obstetrical hemorrhage. Tranexamic acid (TXA) inhibits fibrinolysis and is used routinely to prevent hemorrhage in trauma cases and high risk surgeries. Randomized trials of TXA as a prophylaxis to prevent hemorrhage in cesarean delivery have been small and of mixed quality; however meta-analysis suggests that it is effective.

This study is a randomized placebo-controlled trial of 11,000 women to assess whether tranexamic acid as prophylaxis lowers the risk of postpartum hemorrhage in women undergoing a cesarean delivery.

ELIGIBILITY:
Inclusion Criteria:

1. Scheduled or unscheduled cesarean delivery
2. Singleton or twin gestation

Exclusion Criteria:

1. Age less than 18 years
2. Transfusion or planned transfusion of any blood products during the current admission because the primary outcome is already pre-determined and the need for transfusion will be unrelated to perioperative hemorrhage
3. Recent diagnosis or history of venous thromboembolism or arterial thrombosis because TXA is a risk factor for thromboembolism, and its use is contraindicated
4. Known congenital or acquired thrombophilias, including antiphospholipid antibody syndrome, because of the increased risk of thrombosis
5. Seizure disorder (including eclampsia) because TXA is a GABA receptor antagonist, and its use has been associated with postoperative seizures
6. Serum creatinine 1.2 or higher or on dialysis, with renal disease, or a history of renal insufficiency, because TXA is substantially excreted by the kidney, and impaired renal function may increase the risk of toxic reactions.
7. Sickle cell disease, because of substantial use of perioperative transfusion unrelated to hemorrhage. Sickle cell trait is not an exclusion per se.
8. Autoimmune diseases such as lupus, rheumatoid arthritis, Sjogren's disease, and inflammatory bowel disease because of hypercoagulability and the increased risk of thrombosis or thromboembolism
9. Need for therapeutic dose of anticoagulation before delivery, because the risk of thrombosis may be increased with TXA
10. Treatment with clotting factor concentrates, because the risk of thrombosis may be increased with TXA
11. Presence of frank hematuria, because the risk of ureteral obstruction in those with upper urinary tract bleeding may be increased with TXA
12. Patient refusal of blood products because the primary outcome is then pre-determined
13. Receipt of TXA; or planned or expected use of TXA prophylaxis
14. Active cancer, because of risk of thromboembolism
15. Congestive heart failure requiring treatment, because of risk of thrombosis
16. History of retinal disease, because the risk of central retinal artery or vein obstruction may be increased with TXA
17. Acquired defective color vision or subarachnoid hemorrhage, since TXA is contraindicated
18. Hypersensitivity to TXA or any of the ingredients
19. No hemoglobin result available from the last 4 weeks, since it is necessary to measure the post-operative change in hemoglobin
20. Scheduled cesarean delivery and quota for scheduled deliveries already met. Quotas on the number of scheduled and unscheduled deliveries will be placed to ensure approximately equal distribution of scheduled and unscheduled cesarean deliveries.
21. Participation in this trial in a previous pregnancy. Patients who were screened in a previous pregnancy, but not randomized, may be included.
22. Participating in another intervention study where the primary outcome includes postpartum bleeding or thromboembolism, or the study intervention directly affects postpartum bleeding or thromboembolism
23. Receipt of uterotonics, other than oxytocin, or planned or expected use of uterotonic prophylaxis
24. Symptomatic for COVID-19 infection within 14 days prior to delivery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11000 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2021-07-24 (Actual); Study Completion 2021-10-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Clifton, Ph.D., Principal Investigator — The George Washington University Biostatistics Center; Monica Longo, MD, Study Director — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD); Louis Pacheco, MD, Study Chair — UTMB
Locations (12):
- United States (12):
  - University of Alabama - Birmingham, Birmingham, Alabama
  - Northwestern University-Prentice Hospital, Chicago, Illinois
  - Columbia University, New York, New York
  - University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Case Western Reserve-MetroHealth, Cleveland, Ohio
  - Ohio State University Hospital, Columbus, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Magee Women's Hospital of UPMC, Pittsburgh, Pennsylvania
  - Brown University, Providence, Rhode Island
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas - Houston, Houston, Texas
  - University of Utah Medical Center, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
The dataset will be shared per NIH policy after the completion and publication of the main analyses. Data be will accessible through the NICHD Data and Specimen Hub.

REFERENCES:
- [Background] Hogberg U. The World Health Report 2005: "make every mother and child count" - including Africans. Scand J Public Health. 2005;33(6):409-11. doi: 10.1080/14034940500217037. No abstract available. PMID 16332605
- [Background] Xu J, Kochanek KD, Murphy SL, Tejada-Vera B. Deaths: final data for 2007. Natl Vital Stat Rep. 2010 May;58(19):1-19. PMID 25075874
- [Background] Kwee A, Bots ML, Visser GH, Bruinse HW. Emergency peripartum hysterectomy: A prospective study in The Netherlands. Eur J Obstet Gynecol Reprod Biol. 2006 Feb 1;124(2):187-92. doi: 10.1016/j.ejogrb.2005.06.012. Epub 2005 Jul 18. PMID 16026917
- [Background] Martin JA, Hamilton BE, Osterman MJ, Driscoll AK, Mathews TJ. Births: Final Data for 2015. Natl Vital Stat Rep. 2017 Jan;66(1):1. PMID 28135188
- [Background] Magann EF, Evans S, Hutchinson M, Collins R, Howard BC, Morrison JC. Postpartum hemorrhage after vaginal birth: an analysis of risk factors. South Med J. 2005 Apr;98(4):419-22. doi: 10.1097/01.SMJ.0000152760.34443.86. PMID 15898516
- [Background] Ickx BE. Fluid and blood transfusion management in obstetrics. Eur J Anaesthesiol. 2010 Dec;27(12):1031-5. doi: 10.1097/EJA.0b013e32833c30e3. PMID 20613540
- [Background] Brohi K, Cohen MJ, Davenport RA. Acute coagulopathy of trauma: mechanism, identification and effect. Curr Opin Crit Care. 2007 Dec;13(6):680-5. doi: 10.1097/MCC.0b013e3282f1e78f. PMID 17975390
- [Background] Andersson L, Nilsoon IM, Colleen S, Granstrand B, Melander B. Role of urokinase and tissue activator in sustaining bleeding and the management thereof with EACA and AMCA. Ann N Y Acad Sci. 1968 Jun 28;146(2):642-58. doi: 10.1111/j.1749-6632.1968.tb20322.x. No abstract available. PMID 5254275
- [Background] CRASH-2 trial collaborators; Shakur H, Roberts I, Bautista R, Caballero J, Coats T, Dewan Y, El-Sayed H, Gogichaishvili T, Gupta S, Herrera J, Hunt B, Iribhogbe P, Izurieta M, Khamis H, Komolafe E, Marrero MA, Mejia-Mantilla J, Miranda J, Morales C, Olaomi O, Olldashi F, Perel P, Peto R, Ramana PV, Ravi RR, Yutthakasemsunt S. Effects of tranexamic acid on death, vascular occlusive events, and blood transfusion in trauma patients with significant haemorrhage (CRASH-2): a randomised, placebo-controlled trial. Lancet. 2010 Jul 3;376(9734):23-32. doi: 10.1016/S0140-6736(10)60835-5. Epub 2010 Jun 14. PMID 20554319
- [Background] Oremus K, Sostaric S, Trkulja V, Haspl M. Influence of tranexamic acid on postoperative autologous blood retransfusion in primary total hip and knee arthroplasty: a randomized controlled trial. Transfusion. 2014 Jan;54(1):31-41. doi: 10.1111/trf.12224. Epub 2013 Apr 25. PMID 23614539
- [Background] Makhija N, Sarupria A, Kumar Choudhary S, Das S, Lakshmy R, Kiran U. Comparison of epsilon aminocaproic acid and tranexamic Acid in thoracic aortic surgery: clinical efficacy and safety. J Cardiothorac Vasc Anesth. 2013 Dec;27(6):1201-7. doi: 10.1053/j.jvca.2013.04.003. Epub 2013 Sep 17. PMID 24050855
- [Background] As AK, Hagen P, Webb JB. Tranexamic acid in the management of postpartum haemorrhage. Br J Obstet Gynaecol. 1996 Dec;103(12):1250-1. doi: 10.1111/j.1471-0528.1996.tb09638.x. No abstract available. PMID 8968245
- [Background] Wang HY, Hong SK, Duan Y, Yin HM. Tranexamic acid and blood loss during and after cesarean section: a meta-analysis. J Perinatol. 2015 Oct;35(10):818-25. doi: 10.1038/jp.2015.93. Epub 2015 Jul 30. PMID 26226243
- [Background] Ray I, Bhattacharya R, Chakraborty S, Bagchi C, Mukhopadhyay S. Role of Intravenous Tranexamic Acid on Caesarean Blood Loss: A Prospective Randomised Study. J Obstet Gynaecol India. 2016 Oct;66(Suppl 1):347-52. doi: 10.1007/s13224-016-0915-x. Epub 2016 Jun 25. PMID 27651628
- [Background] Lakshmi SD, Abraham R. Role of Prophylactic Tranexamic Acid in Reducing Blood Loss during Elective Caesarean Section: A Randomized Controlled Study. J Clin Diagn Res. 2016 Dec;10(12):QC17-QC21. doi: 10.7860/JCDR/2016/21702.9050. Epub 2016 Dec 1. PMID 28208943
- [Background] Li C, Gong Y, Dong L, Xie B, Dai Z. Is prophylactic tranexamic acid administration effective and safe for postpartum hemorrhage prevention?: A systematic review and meta-analysis. Medicine (Baltimore). 2017 Jan;96(1):e5653. doi: 10.1097/MD.0000000000005653. PMID 28072700
- [Background] Heesen M, Bohmer J, Klohr S, Rossaint R, van de Velde M, Dudenhausen JW, Straube S. Prophylactic tranexamic acid in parturients at low risk for post-partum haemorrhage: systematic review and meta-analysis. Acta Anaesthesiol Scand. 2014 Oct;58(9):1075-85. doi: 10.1111/aas.12341. Epub 2014 Jul 29. PMID 25069636
- [Background] Shahid A, Khan A. Tranexamic acid in decreasing blood loss during and after caesarean section. J Coll Physicians Surg Pak. 2013 Jul;23(7):459-62. PMID 23823946
- [Background] Ker K, Shakur H, Roberts I. Does tranexamic acid prevent postpartum haemorrhage? A systematic review of randomised controlled trials. BJOG. 2016 Oct;123(11):1745-52. doi: 10.1111/1471-0528.14267. Epub 2016 Aug 24. PMID 27558956
- [Background] Sentilhes L, Lasocki S, Ducloy-Bouthors AS, Deruelle P, Dreyfus M, Perrotin F, Goffinet F, Deneux-Tharaux C. Tranexamic acid for the prevention and treatment of postpartum haemorrhage. Br J Anaesth. 2015 Apr;114(4):576-87. doi: 10.1093/bja/aeu448. Epub 2015 Jan 8. PMID 25571934
- [Background] WOMAN Trial Collaborators. Effect of early tranexamic acid administration on mortality, hysterectomy, and other morbidities in women with post-partum haemorrhage (WOMAN): an international, randomised, double-blind, placebo-controlled trial. Lancet. 2017 May 27;389(10084):2105-2116. doi: 10.1016/S0140-6736(17)30638-4. Epub 2017 Apr 26. PMID 28456509
- [Background] Simonazzi G, Bisulli M, Saccone G, Moro E, Marshall A, Berghella V. Tranexamic acid for preventing postpartum blood loss after cesarean delivery: a systematic review and meta-analysis of randomized controlled trials. Acta Obstet Gynecol Scand. 2016 Jan;95(1):28-37. doi: 10.1111/aogs.12798. Epub 2015 Nov 12. PMID 26698831
- [Background] Wei Z, Liu M. The effectiveness and safety of tranexamic acid in total hip or knee arthroplasty: a meta-analysis of 2720 cases. Transfus Med. 2015 Jun;25(3):151-62. doi: 10.1111/tme.12212. Epub 2015 May 29. PMID 26033447
- [Background] Goswami U, Sarangi S, Gupta S, Babbar S. Comparative evaluation of two doses of tranexamic acid used prophylactically in anemic parturients for lower segment cesarean section: A double-blind randomized case control prospective trial. Saudi J Anaesth. 2013 Oct;7(4):427-31. doi: 10.4103/1658-354X.121077. PMID 24348295
- [Background] Ahmadzia HK, Lockhart EL, Thomas SM, Welsby IJ, Hoffman MR, James AH, Murtha AP, Swamy GK, Grotegut CA. Using antifibrinolytics in the peripartum period - concern for a hypercoagulable effect? J Neonatal Perinatal Med. 2017;10(1):1-7. doi: 10.3233/NPM-16139. PMID 28304315
- [Background] Myles PS, Smith JA, Forbes A, Silbert B, Jayarajah M, Painter T, Cooper DJ, Marasco S, McNeil J, Bussieres JS, McGuinness S, Byrne K, Chan MT, Landoni G, Wallace S; ATACAS Investigators of the ANZCA Clinical Trials Network. Tranexamic Acid in Patients Undergoing Coronary-Artery Surgery. N Engl J Med. 2017 Jan 12;376(2):136-148. doi: 10.1056/NEJMoa1606424. Epub 2016 Oct 23. PMID 27774838
- [Background] Pomp ER, Lenselink AM, Rosendaal FR, Doggen CJ. Pregnancy, the postpartum period and prothrombotic defects: risk of venous thrombosis in the MEGA study. J Thromb Haemost. 2008 Apr;6(4):632-7. doi: 10.1111/j.1538-7836.2008.02921.x. Epub 2008 Jan 31. PMID 18248600
- [Background] Heit JA, Kobbervig CE, James AH, Petterson TM, Bailey KR, Melton LJ 3rd. Trends in the incidence of venous thromboembolism during pregnancy or postpartum: a 30-year population-based study. Ann Intern Med. 2005 Nov 15;143(10):697-706. doi: 10.7326/0003-4819-143-10-200511150-00006. PMID 16287790
- [Background] Pilbrant A, Schannong M, Vessman J. Pharmacokinetics and bioavailability of tranexamic acid. Eur J Clin Pharmacol. 1981;20(1):65-72. doi: 10.1007/BF00554669. PMID 7308275
- [Background] Gilad O, Merlob P, Stahl B, Klinger G. Outcome following tranexamic acid exposure during breastfeeding. Breastfeed Med. 2014 Oct;9(8):407-10. doi: 10.1089/bfm.2014.0027. Epub 2014 Jul 15. PMID 25025926
- [Background] Kamel H, Navi BB, Sriram N, Hovsepian DA, Devereux RB, Elkind MS. Risk of a thrombotic event after the 6-week postpartum period. N Engl J Med. 2014 Apr 3;370(14):1307-15. doi: 10.1056/NEJMoa1311485. Epub 2014 Feb 13. PMID 24524551
- [Background] Novikova N, Hofmeyr GJ, Cluver C. Tranexamic acid for preventing postpartum haemorrhage. Cochrane Database Syst Rev. 2015 Jun 16;2015(6):CD007872. doi: 10.1002/14651858.CD007872.pub3. PMID 26079202
- [Derived] Pacheco LD, Clifton RG, Saade GR, Weiner SJ, Parry S, Thorp JM Jr, Longo M, Salazar A, Dalton W, Tita ATN, Gyamfi-Bannerman C, Chauhan SP, Metz TD, Rood K, Rouse DJ, Bailit JL, Grobman WA, Simhan HN, Macones GA; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Tranexamic Acid to Prevent Obstetrical Hemorrhage after Cesarean Delivery. N Engl J Med. 2023 Apr 13;388(15):1365-1375. doi: 10.1056/NEJMoa2207419. PMID 37043652

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We conducted this multicenter, randomized, controlled, double blinded trial at 31 hospitals. From March 2018 through July 2021, a total of 84,062 patients underwent screening for randomization. Of the 39,488 eligible patients, 11,000 provided informed consent and were randomized
Pre-assignment Details: No participants were excluded after enrollment but before assignment to groups.
Period: Overall Study
Arm/Group | Tranexamic Acid | Placebo
Started | 5529 | 5471
Completed | 5529 | 5471
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Of 5529 participants, 4 were enrolled in the study for a second pregnancy in the tranexamic acid group and out of 5471 participants, 1 was enrolled for a second pregnancy in the placebo group. Only the first pregnancy was included in the analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tranexamic Acid | Placebo | Total
Number analyzed (Participants) | 5525 | 5470 | 10995
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.1 (5.8) | 30.1 (5.8) | 30.1 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5525 | 5470 | 10995
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 2170 | 2159 | 4329
  Non-Hispanic Black | 1334 | 1310 | 2644
  Hispanic | 1636 | 1642 | 3278
  Asian | 218 | 193 | 411
  Other, unknown, or more than one race or ethnic group | 167 | 166 | 333
Preoperative Hemoglobin <8g/dL [Count of Participants; unit: Participants] — Population: Values are unavailable for 2 participants in the TXA group and 6 participants in the placebo group.
  Participants
    number analyzed (Participants) | 5523 | 5464 | 10987
    (all) | 10 | 26 | 36

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Maternal Death or Transfusion of Packed Red Blood Cells
Description: Participants were monitored from delivery until hospital discharge or 7 days after delivery (postpartum), whichever is sooner. This is the number of mothers who died for any reason, or had a blood transfusion of 1 or more units (of packed red blood cells, including whole blood or cell saver).
Time Frame: by hospital discharge or by 7 days postpartum, whichever is sooner
Population: Of 5529 participants, 4 were enrolled in the study for a second pregnancy in the tranexamic acid group and out of 5471 participants, 1 was enrolled for a second pregnancy in the placebo group. Since participants were only permitted to be enrolled in the study one time, only the first pregnancy was included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Tranexamic Acid | Placebo
Number analyzed (Participants) | 5525 | 5470
Participants | 201 | 233
Statistical Analysis 1: Comparison: Tranexamic Acid; Test type: Superiority — Model included treatment and preoperative hemoglobin level <8 g/dL (yes/no) as covariates. We estimated that a total sample size of 11,000 participants (5,500 per group) would achieve 85% power to detect a 33% lower incidence of the primary outcome (1.67%) in the TXA group, at a type I error rate (two-sided) of 5%; p = 0.19, Other (Log-binomial regression model) — Following two interim analyses, a two-tailed P value of less than 0.047 was considered to indicate statistical significance; Risk Ratio (RR) = 0.89, 95.26% CI 2-sided [0.74 to 1.07]

2. Secondary Outcome: Number of Participants With Estimated Blood Loss Greater Than 1 Liter During Delivery
Description: [Major secondary outcome] The surgeon or anesthesiologist estimated the blood loss during the delivery in milliliters, which was recorded in the anesthesia record and/or operative report
Time Frame: From skin incision to transfer from operating room, average of 1 hour
Population: All participants for which blood loss data is available in the anesthesia record and/or operative report are included. Additionally, 5 enrolled for a second pregnancy (4 in the tranexamic acid group and 1 in the placebo group) only included the result from the first enrolled pregnancy (when available) since participants were only permitted to be enrolled in the study one time.
Measure: Count of Participants; unit: Participants
Arm/Group | Tranexamic Acid | Placebo
Number analyzed (Participants) | 4641 | 4573
Participants | 339 | 368

3. Secondary Outcome: Number of Mothers Who Died or Had Thromboembolic Events (Venous or Arterial), Ischemic Stroke, Myocardial Infarction, New-onset Seizure Activity, or Were Admitted to the Intensive Care Unit for More Than 24 Hours
Time Frame: within 6 weeks postpartum
Population: Participants who received study medication are included according to the treatment received; only those with follow-up through 6 weeks postpartum are included. Additionally, 5 enrolled for a second pregnancy (4 in the tranexamic acid group and 1 in the placebo group) only included the result from the first enrolled pregnancy (when available) since participants were only permitted to be enrolled in the study one time.
Measure: Count of Participants; unit: Participants
Arm/Group | Tranexamic Acid | Placebo
Number analyzed (Participants) | 5069 | 4996
Participants | 35 | 32

4. Secondary Outcome: Number of Participants Who Were Transfused With Other Blood Products
Description: This is the number of mothers who received during the first 7 days after delivery a transfusion of 1 or more units of fresh frozen plasma, cryoprecipitate, or platelets, or received any factor concentrates
Time Frame: within 7 days postpartum
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Tranexamic Acid | Placebo
Number analyzed (Participants) | 5525 | 5470
Participants | 29 | 31

5. Secondary Outcome: Number of Participants Who Were Transfused With 4 or More Units of Packed Red Blood Cells
Description: Participants were categorized according to the amount of packed red blood cells or whole blood transfused, either as 0 to 3 units, or 4 or more units
Time Frame: within 7 days postpartum
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Tranexamic Acid | Placebo
Number analyzed (Participants) | 5525 | 5470
Participants | 20 | 19

6. Secondary Outcome: Number of Participants With a Thromboembolic Event (Venous or Arterial), Ischemic Stroke, or Myocardial Infarction
Description: [Key secondary outcome] This is the number of mothers who experienced a thromboembolic event, ischemic stroke, or myocardial infarction during the 6 weeks after delivery.
Time Frame: within 6 weeks postpartum
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Tranexamic Acid | Placebo
Number analyzed (Participants) | 5069 | 4996
Participants | 12 | 13

7. Secondary Outcome: Number of Participants With Seizure Activity That Was Not Seen Prior to Study Enrollment
Description: This is the number of mothers who experienced seizure activity, confirmed by central review, whose onset is after enrollment
Time Frame: within 6 weeks postpartum
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Tranexamic Acid | Placebo
Number analyzed (Participants) | 5069 | 4996
Participants | 2 | 0

8. Secondary Outcome: Number of Participants With Postpartum Infectious Complications
Description: [Key Secondary Outcome] This is the number of mothers who experienced any of the following infectious complications in the 6 weeks after delivery: endometritis, surgical site infection, pelvic abscess
Time Frame: within 6 weeks postpartum
Population: Only those with follow-up through 6 weeks postpartum are included. Additionally, 5 enrolled for a second pregnancy (4 in the tranexamic acid group and 1 in the placebo group) only included the result from the first enrolled pregnancy (when available) since participants were only permitted to be enrolled in the study one time.
Measure: Count of Participants; unit: Participants
Arm/Group | Tranexamic Acid | Placebo
Number analyzed (Participants) | 5080 | 5009
Participants | 162 | 125

9. Secondary Outcome: Number of Participants Who Were Treated With Uterotonics Other Than Oxytocin
Description: This is the number of mothers who were treated with uterotonics such as prostaglandins or methergine, but excluding oxytocin, from delivery through 48 hours after delivery.
Time Frame: within 48 hours postpartum
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Tranexamic Acid | Placebo
Number analyzed (Participants) | 5525 | 5470
Participants | 649 | 732

10. Secondary Outcome: Number of Participants Who Received Surgical or Radiologic Interventions to Control Bleeding and Related Complications
Description: This is the number of mothers who required any of the following types of surgical procedures to control bleeding: laparotomy, evacuation of hematoma, hysterectomy, uterine packing, intrauterine balloon tamponade, interventional radiology
Time Frame: within 7 days postpartum
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Tranexamic Acid | Placebo
Number analyzed (Participants) | 5525 | 5470
Participants | 233 | 231

11. Secondary Outcome: Change in Hemoglobin
Description: [Key secondary outcome] Change in hemoglobin from the most recent measured before delivery to lowest measured in the 48 hours after delivery
Time Frame: from 4 weeks before delivery to 48 hours postpartum
Population: Only those with both hemoglobin measurements before and after delivery are included. Additionally, 5 enrolled for a second pregnancy (4 in the tranexamic acid group and 1 in the placebo group) only included the result from the first enrolled pregnancy (when available) since participants were only permitted to be enrolled in the study one time.
Measure: Mean (Standard Error); unit: grams per deciliter
Arm/Group | Tranexamic Acid | Placebo
Number analyzed (Participants) | 5224 | 5201
grams per deciliter | -1.8 (1.1) | -1.9 (1.1)

12. Secondary Outcome: Number of Participants Who Received Open Label TXA or Other Antifibrinolytic
Description: This is the number of mothers who were treated with any amount of open-label TXA (not blinded study drug) or another antifibrinolytic (eg., Amicar)
Time Frame: within 7 days postpartum
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Tranexamic Acid | Placebo
Number analyzed (Participants) | 5525 | 5470
Participants | 108 | 109

13. Secondary Outcome: Length of Stay
Description: Mother's length of stay from delivery to discharge
Time Frame: Until hospital discharge, an average of 3 days
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Tranexamic Acid | Placebo
Number analyzed (Participants) | 5525 | 5470
days | 3 [2 to 3] | 3 [2 to 3]

14. Secondary Outcome: Number of Participants Who Received Treatments and Interventions in Response to Bleeding and Related Complications
Description: [Key secondary outcome] This is the number of mothers who received treatments and interventions to control bleeding such as: uterotonics such as prostaglandins or methergine, but excluding oxytocin; open label TXA or other antifibrinolytics; transfusion of 1 or more units of fresh frozen plasma, cryoprecipitate, or platelets or administration of any factor concentrates; laparotomy, evacuation of hematoma, hysterectomy, uterine packing, intrauterine balloon tamponade, interventional radiology
Time Frame: within 7 days postpartum
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Tranexamic Acid | Placebo
Number analyzed (Participants) | 5525 | 5470
Participants | 892 | 986

ADVERSE EVENTS:
Time Frame: Within 6 weeks postpartum
Description: All-cause mortality includes maternal, fetal, and neonatal deaths. Unless otherwise specified, all other adverse events are for the pregnant or postpartum participant.
Arm/Group | Tranexamic Acid | Placebo
All-Cause Mortality (participants affected / at risk) | 26/5529 | 32/5471
Serious Adverse Events (participants affected / at risk) | 82/5529 | 70/5471
Other Adverse Events (participants affected / at risk) | 593/5529 | 647/5471
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tranexamic Acid (N=5529) | Placebo (N=5471)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiomegaly (Cardiac disorders) | 0 (0) | 1 (1)
Heart failure/ Cardiomyopathy (Cardiac disorders) | 4 (4) | 5 (5)
Pericardial Effusion (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea/vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 3 (3) | 1 (1)
Gastric Ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1)
Small bowel obstruction (Gastrointestinal disorders) | 2 (2) | 1 (1)
fever (General disorders) | 1 (1) | 0 (0)
neonatal drug withdrawal (General disorders) | 1 (1) | 0 (0)
cholelithiasis/ cholecystitis (Hepatobiliary disorders) | 2 (2) | 5 (5)
Anaphylaxis (Immune system disorders) | 1 (1) | 0 (0)
Myasthenia gravis (Immune system disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Necrotizing soft tissue infection (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 1 (1)
respiratory infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 5 (5) | 5 (5)
Septic Thrombophlebitis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
other undefined infection (Infections and infestations) | 0 (0) | 1 (1)
Wound dehiscence, seroma, hematoma, or cellulitis (Injury, poisoning and procedural complications) | 4 (4) | 3 (3)
Neonatal vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Bell's Palsy (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Spinal headache (Nervous system disorders) | 1 (1) | 0 (0)
Neonatal Seizure/stroke (Nervous system disorders) | 2 (2) | 0 (0)
Neonatal cerebral arterial or venous infarction (Nervous system disorders) | 1 (1) | 1 (1)
Neonatal hypotonia (Nervous system disorders) | 0 (0) | 1 (1)
Preeclampsia and associated complications (Pregnancy, puerperium and perinatal conditions) | 28 (28) | 22 (22)
Depression (Psychiatric disorders) | 0 (0) | 2 (2)
Pyschosis (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Mastitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Air embolism (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
Neonatal thrombosis or occlusion (Vascular disorders) | 2 (2) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 1.0% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tranexamic Acid (N=5529) | Placebo (N=5471)
Nausea (Gastrointestinal disorders) | 363 | 404
Vomiting (Gastrointestinal disorders) | 266 | 273
Dizziness (Nervous system disorders) | 157 | 186
Urticaria or dermatitis (Skin and subcutaneous tissue disorders) | 63 | 72

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-04-08): https://cdn.clinicaltrials.gov/large-docs/91/NCT03364491/Prot_SAP_ICF_000.pdf